CLINICAL TRIAL: NCT04028778
Title: A Multicenter, Randomized, Double-Blind Study of Gefitinib in Combination With Anlotinib or Placebo in Previously Untreated Patients With EGFR Mutation-Positive Advanced Non-Small-Cell Lung Cancer
Brief Title: Gefitinib in Combination With Anlotinib or Placebo in Previously Untreated EGFR-mutant NSCLC
Acronym: FL-ALTER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-FXY-134-内科
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Blind Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gefitinib + Anlotinib (Experimental): Patients will be treated with Gefitinib 250mg, p.o., qd and anlotinib hydrochloride capsule 12mg, p.o., qd, D1-D14; take on an empty stomach (take at the same time every day as possible), every 3 weeks for a cycle.
  Interventions: Drug: Gefitinib; Drug: Anlotinib Hydrochloride
- Gefitinib + Placebo (Placebo Comparator): Patients will be treated with Gefitinib 250mg, p.o., qd and placebo to simulate anlotinib hydrochloride capsule 12mg, p.o., qd, D1-D14; take on an empty stomach (take at the same time every day as possible), every 3 weeks for a cycle
  Interventions: Drug: Gefitinib; Other: Placebo

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg, p.o., qd, D1-D21; 3 weeks one cycle.
  Other Names: Iressa
Drug: Anlotinib Hydrochloride — Anlotinib hydrochloride capsule 12mg, p.o., qd, D1-D14; 3 weeks one cycle.
  Arms: Gefitinib + Anlotinib
Other: Placebo — Placebo simulating anlotinib hydrochloride capsule 12mg, p.o., qd, D1-D14; 3 weeks one cycle.
  Arms: Gefitinib + Placebo

SUMMARY:
Gefitinib is currently the standard-of-care for patients with activating-EGFR mutant advanced non-small cell lung cancer (NSCLC). However, ~30-40% patients are still nonresponsive, and experience significantly varying duration of response and survival rate. Anlotinib is an efficient multi-target tyrosine kinase inhibitor (TKI) that effectively block the migration and proliferation of endothelial cells and reduce tumor microvascular density by targeting VEGFRs, FGFRs, PDGFRs. It has been proved to be safe and effective in advanced lung cancer after second-line standard chemotherapy failure, which can significantly extend the survival of patients and approves as a third-line treatment for advanced NSCLC. Here, we prepared to evaluate whether the combination of gefitinb and anlotinib can preferably improved survival of untreated NSCLC with EGFR activating mutation.

ELIGIBILITY:
Inclusion Criteria:

* 1.≥ 18 and ≤ 75 years of age
* 2.Eastern Cooperative Oncology Group(ECOG)performance scale 0 - 1.
* 3.Life expectancy of more than 3 weeks
* 4.Histologically confirmed，locally advanced and/or metastatic non-squamous NSCLC of stage IIIB (unsuitable for radiotherapy) or IV or recurrent NSCLC with measurable lesion/ according to RECIST 1.1 which has not received radiotherapy or cryotherapy.
* 5.Documented evidence of tumor harboring an activating EGFR mutation (exon19 del and L858R)
* 6.None previous chemotherapy or targeted therapy. NOTE: neoadjuvant and/or adjuvant therapy is allowed which is completed before 6 months
* 7.Prior radiation therapy is allowed if: 25% or less of total bone marrow had been irradiated,pelvis and chest had not been irradiated; at least 4 weeks have elapsed from the completion of radiation treatment, and the acute toxicity from radiation treatment had been recover; irradiated lesion is not including measurable lesions unless documented progress after radiation.
* 8.Adequate hepatic, renal, heart, and hematologic functions (Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 100×109/L, Hemoglobin(HB) ≥ 100 g/L, total bilirubin within 1.5×the upper limit of normal(ULN), and serum transaminase≤2.5×the Upper Limit Of Normal(ULN), serum creatine ≤ 1 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥ 50ml/min
* 9.For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
* 10.Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* 1.small cell lung cancer (including small cell and non-small cell mixed lung cancer)
* 2.Symptomatic brain metastases (Patients who have no symptoms and is not needed to receive therapy before 21 days may participate in this trial, but need to be confirmed by MRI\CT or venography that no hematencephalon symptom)
* 3.Radiologically documented evidence of tumor lesions from large vessels ≤ 5mm or major blood vessel invasion or encasement by cancer; Obvious cavity or necrosis formed in the tumor.
* 4. hypertensive patients are in the combination therapy of two or more antihypertensive drugs.
* 5.patients with positive T790M mutation by Gene detection.
* 6.Patients who suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
* 7.History of pulmonary interstitial diseases or concurrent pulmonary interstitial diseases.
* 8.Coagulation disfunction（INR>1.5 or PT>Upper Limit Of Normal(ULN)+4s or Activated Partial Thromboplastin Time (APTT) >1.5 Upper Limit Of Normal(ULN)）, hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation
* 9.Daily hemoptysis up to two teaspoons or more before enrollment
* 10.History of clinically relevant major bleeding event=<3 months (e.g. gastrointestinal hemorrhage, Hemorrhagic acne， bleeding gastric ulcer, occult blood test ≥ (++), and vasculitis ;
* 11.Within 12 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack(TIA), hematencephalon, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* 12.Known inherited and acquired hemorrhagic and thromboplastic possibility (such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.)
* 13.Long-term untreated wounds or fractures（in addition to tumor-induced pathological fractures）
* 14.Within 4 weeks of major surgery and/or injures, fractures , ulceration
* 15.Significant factors that influence the ingestion and absorption of medicine, (e.g. unable swallow, chronic diarrhea and intestinal obstruction);
* 16.History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 6 months.
* 17.Urine protein≥++, and 24h urine protein quantitation≥1.0g;
* 18.Symptomatic serous effusion requiring treatment .(including hydrothorax, ascites, hydropericardium);
* 19.Active infection need antimicrobial treatments（such as antibiotics and antiviral drugs should be used, excluding anti-hepatitis B treatment and antifungal therapy. ）
* 20.History of psychiatric drugs abuse and not be abstinent, or dysphrenia
* 21.Less than 4 weeks from the last clinical trial
* 22.History or concomitant other malignancy except cured basal cell skin cancer, or carcinoma in situ of the cervix, or superficial bladder cancer;
* 23.Administration of strong/potent cytochrome P450 (CYP)3A4 inhibitors within 7 days, or inducers within 12 days;
* 24.Pregnant or breastfeeding women；patients who have fertility are unwilling or unable to take effective contraceptive measures;
* 25.Other conditions regimented at investigators' discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | Approximately 2 Years
  Progression-Free Survival (PFS) as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1)

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 5 Years
  OS was defined as the time from the date of randomization to the date of death due to any cause.
Percentage of Participants With Objective Response (Partial Response [PR] Plus Complete Response [CR]), as Assessed Using RECIST v.1.1 | Approximately 2 Years
  PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions).
Percentage of Participants With Clinical Benefit, as Assessed According to RECIST v1.1 | Approximately 2 Years
  Clinical benefit was defined as objective response (PR+CR), or no disease progression lasting for more than or equal to (>/=) 24 weeks since randomization. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions). Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.
Duration of Objective Response, as Assessed by Investigator Using RECIST v1.1 | Approximately 2 Years
  Duration of objective response: the time from the first tumor assessment that supported the participant's objective response (CR or PR, whichever was first recorded) to first documented disease progression or death due to any cause, whichever occurred first. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Disease progression: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression.

OTHER OUTCOMES:
Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Score | Approximately 2 Years
  The EORTC QLQ-C30 consists of 30 questions that comprise aspects of participant's functioning assessment (physical, emotional, role, cognitive, and social); symptom scales (fatigue; nausea, vomiting, and pain; the global health/quality of life [QoL]); and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties), within a recall period of "the past week." Most questions used a 4-point scale (1=Not at all to 4=Very much; two questions used a 7-point scale (1=Very poor to 7=Excellent). Scores were averaged and transformed to a 0-100 scale; a higher score for Global Qol/functional scales=better level of functioning; a higher score for symptom scale=greater degree of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University (CCSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou HQ, Zhang YX, Chen G, Yu QT, Zhang H, Wu GW, Wu D, Lin YC, Zhu JF, Chen JH, Hu XH, Lan B, Zhou ZQ, Lin HF, Wang ZB, Lei XL, Pan SM, Chen LM, Zhang J, Kong TD, Yao JC, Zheng X, Li F, Zhang L, Fang WF. Gefitinib (an EGFR tyrosine kinase inhibitor) plus anlotinib (an multikinase inhibitor) for untreated, EGFR-mutated, advanced non-small cell lung cancer (FL-ALTER): a multicenter phase III trial. Signal Transduct Target Ther. 2024 Aug 13;9(1):215. doi: 10.1038/s41392-024-01927-9. PMID 39134529